CLINICAL TRIAL: NCT05278169
Title: Central Serous Chorioretinopathy Registry and Pachychoroid Observation and Natural History Study
Acronym: CSCR POOH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Danny Siu-Chun NG, Associate Professor, Chinese University of Hong Kong
Other Study IDs: CSCR POOH
Record Dates: First submitted 2022-01-17; First posted 2022-03-14 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Central Serous Chorioretinopathy; Pachychoroid; Optical Coherence Tomography
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — A 10 mL blood sample will be drawn by venipuncture during the first (baseline) visit for genetics analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives:

1. To conduct a Natural History Observation Study to characterize the clinical features and progression of Central Serous Chorioretinopathy (CSCR) from the earliest to the vision-threatening stages.
2. Collect genetic samples of affected individuals and their families to establish whether there is a genetic basis for the disease.
3. To create a Registry of patients affected by CSCR who may agree to be contacted for inclusion in future clinical trials.
4. To determine the incidence and risk factors for progression of pachychoroid phenotypes identified from the unaffected fellow eyes of CSCR patients.

Design and subjects:

Observation, non-interventional study with prospective follow-up for 2 years. The study aims to enroll 350 patients with CSCR (100 from Hong Kong Eye Hospital, 80 from Prince of Wales Hospital and Alice Ho Miu Ling Nethersole Hospital, and 170 from Chinese University of Hong Kong (CUHK) Eye Centre at Hong Kong Eye Hospital).

Study instruments:

Functional tests include visual acuity and microperimetry. Retinal imaging with non-invasive ultra-widefield colour fundus camera, fundus autofluorescence (FAF) and optical coherence tomography (OCT). Questionnaires for risk factor profiling and quality of life assessment. Blood specimen will be collected for genetic testing if found to have a clinical diagnosis of CSCR as determined at CUHK Eye Centre at Hong Kong Eye Hospital.

Main outcome measures:

The primary outcome will be longitudinal alteration of retinal pigment epithelium defects on FAF, spectral domain (SD) OCT and infrared imaging. The secondary outcomes are: 1) progressive attenuation of outer nuclear layer (ONL), external limiting membrane (ELM) and ellipsoid zone (EZ) on SD OCT, 2) longitudinal changes of subfoveal choroidal thickness on swept source (SS) OCT, 3) incidence and onset of intraretinal cysts, 4) incidence and onset of type 1 choroidal neovascularization, 5) rate of choriocapillaris non- perfusion on SS OCT angiography (OCTA), 6) rate of loss of retinal sensitivity using microperimetry tests, 7) rate of visual acuity loss, 8) epidemiology of risk factors associated with CSCR, 9) identification of genes and the genetic variants that are associated with susceptibility to CSCR and 10) documentation of the clinical course of serous retinal detachment recurrence(s), persistence and resolution.

DETAILED DESCRIPTION:
Significance and Applications of Study Results:

I) The proposed study will determine comprehensive clinical characterization of a large cohort of 350 CSCR patients with novel, non-invasive imaging techniques to examine the ultrastructure of the choroid and retina to detect subtle changes that are not visible through routine eye check and conventional fundoscopy examination.

II) To understand the pathophysiology of CSCR through studying ultrastructural changes of chorioretina and genotypes.

III) Longitudinal data from this study will determine CSCR progression risks and treatment outcomes. Our large CSCR database will be a unique, large cohort study with robust clinical and molecular characterizations. This knowledge could help to develop realistic and effective diagnostic tests and individualized treatments for CSCR, and aid in the design of future clinical trials.

Data analysis:

Statistical analyses will be conducted using standard statistical software (SPSS, STATA). The investigators will use a variety of statistical techniques for analysis. Unless otherwise specified, all statistical tests will be two-sided with a 0.05 level of significance. All confidence intervals will be two-sided with 95% confidence level. Categorical variables will be presented as the number and percentage of patients in each category. Continuous variables will be summarized using descriptive statistics such as n, mean, standard deviation, median, minimum, and maximum.

Descriptive statistics will be provided for patient demographics and baseline characteristics. Other relevant baseline information will be listed and summarized as appropriate with descriptive statistics.

An independent committee will review the data and safety of the study. Adequate records will be maintained and made available for audit / inspection. All study documents will be kept for a period of at least three years after study closure.

Significant Differences from Usual Management:

1. The study is a prospective natural history observation study and the protocol requires a total of 5 visits (in addition to routine care) to the CUHK Eye Centre at Hong Kong Eye Hospital for a duration of 2 years.
2. Blood taking will only be performed during the first (baseline) visit for genetic study.

Methods:

For Visit 1 (Baseline, Month 0):

1. Demography and Past medical history (1.1. Medical history, 1.2. Drugs history, 1.3. Blood pressure (BP) and Body-mass index (BMI) measurements, 1.4. Previous fluorescein and indocyanine green angiography images (if available) will be reviewed)
2. Visual function, intraocular pressure and ocular biometry (2.1. Best corrected visual acuity, 2.2. Autorefraction, 2.3. Axial length measurement, 2.4. Fundus Autofluorescence, 2.5. Macular Spectral Domain Optical Coherence Tomography (SD-OCT) 2.6. Ultra-widefield color fundus photography and autofluorescence, 2.7. Macular Swept Source Optical Coherence Tomography (SS-OCT), 2.8. OCT angiography, 2.9. Microperimetry)
3. Sleep quality, mood and quality of life questionnaires (3.1. Morningness and Eveningness Questionnaire, 3.2. Pittsburgh Sleep Quality Index (PSQI), 3.3. Insomnia Severity Index (ISI), 3.4. Epworth Sleepiness Scale (ESS), 3.5. General Anxiety Disorder-7 (GAD-7) and Patient Health Questionnaire-9 (PHQ-9) questionnaires, 3.6. National Eye Institute Visual Functioning Questionnaire - 25 (NEI-VFQ-25) quality of life questionnaire)
4. Blood taking for genetic study

For Visit 2 (Month 6) to Visit 5 (Months 24):

1.1 to 1.4 will be reviewed for any updates. The eye investigations that will be repeated are: 2.1, 2.4 - 2.9 The questionnaires that will be repeated are: 3.5 - 3.6 (only during Visits 3 and 5)

ELIGIBILITY:
Inclusion Criteria:

* Presence or evidence of prior serous retinal detachment documented on OCT involving the posterior pole unrelated to another disease process.
* At least 1 area of retinal pigment epithelium (RPE) alteration on FAF, SD-OCT, or infrared imaging.
* Subfoveal choroidal thickness (SFCT) of 300μm or more on SD enhanced depth imaging (EDI) OCT or SS-OCT for at least one eye.
* Patient 18 years or older.
* Willing to undergo pupil dilation, and protocol-required procedures for both eyes.

Exclusion Criteria:

* Other maculopathy on clinical examination such as age-related macular degeneration (AMD).
* Media opacity such as cataract that could interfere with adequate acquisition of fundal images.
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to enrol a total of 350 patients with CSCR, of which:
  * 170 subjects from a previous cross-sectional observation study titled 'The Association of Sleep Disturbances and Maculopathy' (IRB / REC No.: 2018.158) at the CUHK Eye Centre.
  * An addition of 180 subjects will be recruited during the proposed study duration. Of the 180 new recruits, 100 will be recruited from Hong Kong Eye Hospital and CUHK Eye Centre.The remaining 80 subjects will be recruited from Department of Ophthalmology and Visual Sciences, Prince of Wales Hospital and Alice Ho Miu Ling Nethersole Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal change of retinal pigment epithelium defects on Fundus Autofluorescence (FAF) from baseline and between visits. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Fundus Autofluorescence - performed using Spectralis (Heidelberg Engineering, Heidelberg, Germany) to acquire 35 degree and 55 degree image centred on the fovea.
Longitudinal change of retinal pigment epithelium defects on Spectral Domain Optical Coherence Tomography (SD-OCT) from baseline and between visits. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Macular Spectral Domain Optical Coherence Tomography (SD-OCT) - performed using Spectralis (Heidelberg Engineering, Heidelberg, Germany) to acquire a 6x6 mm cube comprising of 97 retinal scans centred on the fovea.
Longitudinal change of retinal pigment epithelium defects on infrared imaging from baseline and between visits. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Ultra-widefield color fundus photography and autofluorescence (Optos PLC, Dunfermline, UK) - performed to capture 240 degree image centred on the fovea.

SECONDARY OUTCOMES:
Progressive attenuation of outer nuclear layer (ONL), external limiting membrane (ELM) and ellipsoid zone (EZ) on SD-OCT. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Macular Spectral Domain Optical Coherence Tomography (SD-OCT) - performed using Spectralis (Heidelberg Engineering, Heidelberg, Germany) to acquire a 6x6 mm cube comprising of 97 retinal scans centred on the fovea.
Changes of subfoveal choroidal thickness on swept source optical coherence tomography (SS-OCT). | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Macular Swept Source Optical Coherence Tomography (SS-OCT) - performed using Triton Deep Range Imaging OCT (Topcon Corp., Tokyo, Japan) to acquire 12 raster radial lines (300 x 50), 1 clock hour apart and centered on the fovea, with 16 frames averaged in each B-scan. Each scan is 12mm in length. Bruch's membrane and choroidal-scleral interface (CSI) were delineated with the machine's built-in autosegmentation software, with manual adjustments if necessary. Subfoveal choroidal thickness (SFCT) is defined as the distance from the Bruch's membrane and CSI and was automatically measured by built-in caliper at the fovea.
Incidence of intraretinal cysts. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Determined by retinal imaging with non-invasive ultra-widefield colour fundus camera, fundus autofluorescence (FAF) and optical coherence tomography (OCT).
Onset of intraretinal cysts. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Determined by retinal imaging with non-invasive ultra-widefield colour fundus camera, fundus autofluorescence (FAF) and optical coherence tomography (OCT).
Incidence of type 1 choroidal neovascularization. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Determined by retinal imaging with non-invasive ultra-widefield colour fundus camera, fundus autofluorescence (FAF) and optical coherence tomography (OCT).
Onset of type 1 choroidal neovascularization. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Determined by retinal imaging with non-invasive ultra-widefield colour fundus camera, fundus autofluorescence (FAF) and optical coherence tomography (OCT).
Changes of choriocapillaris non-perfusion on SS OCT angiography (OCTA). | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  OCT angiography (OCTA) - performed using the Triton Deep Range Imaging OCT (Topcon Corp., Tokyo, Japan) to acquire 6mm macular cube in resolution of 512x512 and 3D OCT image. Each eye will be scanned in duplicate (3 times) so that averaging can be performed for choriocapillaris flow void quantification.
Changes of retinal sensitivity using microperimetry tests. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Microperimetry (MAIA, Italy) for macular function and sensitivity assessment.
Visual acuity changes. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Best corrected visual acuity (ETDRS chart letter score).
Epidemiological association of medical history with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Detailed survey will be conducted on smoking status and medical history including hypertension, coronary heart disease, cerebrovascular disease, erectile dysfunction, Helicobacter pylori infection, peptic ulcer, gastroesophageal reflux, autoimmune diseases, organ transplant, pregnancy, eczema, endocrine diseases such as Cushing syndrome, anxiety and depression.
Epidemiological association of use of oral corticosteroids with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of use of intravenous corticosteroids with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of use of intravitreal corticosteroids with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of use of periocular corticosteroids with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of use of intranasal corticosteroids with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of use of intra-articular corticosteroids with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of use of epidural corticosteroids with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of use of dermal corticosteroids with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of use of antacids with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of use of antihistamines with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of use of nasal sprays that contain pseudoephedrine and oxymetazoline with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of use of phosphodiesterase-5 inhibitors with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Phosphodiesterase-5 inhibitors such as sildenafil.
Epidemiological association of blood pressure (BP) with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of body-mass index (BMI) with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of previous findings in fluorescein and indocyanine green angiography images with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
Epidemiological association of best corrected visual acuity with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Best corrected visual acuity as measured by ETDRS chart letter score.
Epidemiological association of autorefraction with CSCR. | At baseline (Month 0).
Epidemiological association of axial length measurement with CSCR. | At baseline (Month 0).
  Axial length measurement as measured by IOL-Master (Zeiss, Germany).
Epidemiological association of findings in Fundus Autofluorescence with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Fundus Autofluorescence will be performed using Spectralis (Heidelberg Engineering, Heidelberg, Germany) to acquire 35 degree and 55 degree image centred on the fovea.
Epidemiological association of findings in Macular Spectral Domain Optical Coherence Tomography (SD-OCT) with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Macular Spectral Domain Optical Coherence Tomography (SD-OCT) will be performed using Spectralis (Heidelberg Engineering, Heidelberg, Germany) to acquire a 6x6 mm cube comprising of 97 retinal scans centred on the fovea.
Epidemiological association of findings in ultra-widefield color fundus photography and autofluorescence with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Ultra-widefield color fundus photography and autofluorescence (Optos PLC, Dunfermline, UK) will be performed to capture 240 degree image centred on the fovea.
Epidemiological association of findings in Macular Swept Source Optical Coherence Tomography (SS-OCT) with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Macular Swept Source Optical Coherence Tomography (SS-OCT) will be performed using Triton Deep Range Imaging OCT (Topcon Corp., Tokyo, Japan) to acquire 12 raster radial lines (300 x 50), 1 clock hour apart and centered on the fovea, with 16 frames averaged in each B-scan. Each scan is 12mm in length. Bruch's membrane and choroidal-scleral interface (CSI) were delineated with the machine's built-in autosegmentation software, with manual adjustments if necessary. Subfoveal choroidal thickness (SFCT) is defined as the distance from the Bruch's membrane and CSI and was automatically measured by built-in caliper at the fovea.
Epidemiological association of findings in OCT angiography with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  OCT angiography will be performed using the Triton Deep Range Imaging OCT (Topcon Corp., Tokyo, Japan) to acquire 6mm macular cube in resolution of 512x512 and 3D OCT image. Each eye will be scanned in duplicate (3 times) so that averaging can be performed for choriocapillaris flow void quantification.
Epidemiological association of findings in microperimetry with CSCR. | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Microperimetry (MAIA, Italy) will be preformed for macular function and sensitivity assessment.
Epidemiological association of morningness - eveningness choronotype with CSCR. | At baseline (Month 0).
  The brief version of the Morningness- Eveningness Questionnaire, which has been validated in Chinese population with satisfactory psychometric properties, will be employed to measure the chronotype.
Epidemiological association of sleep quality with CSCR. | At baseline (Month 0).
  Pittsburgh Sleep Quality Index (PSQI) for evaluating one's overall sleep quality and the severity of insomnia symptoms, respectively. Minimum Score: 0. Maximum Score: 21. A higher score means a worse sleep quality.
Epidemiological association of severity of insomnia with CSCR. | At baseline (Month 0).
  Insomnia Severity Index (ISI) for evaluating one's overall sleep quality and the severity of insomnia symptoms, respectively. Minimum Score: 0. Maximum Score: 28. A higher score means a higher severity of insomnia.
Epidemiological association of excessive daytime sleepiness with CSCR. | At baseline (Month 0).
  Epworth Sleepiness Scale (ESS): ESS will be also employed to measures excessive daytime sleepiness in our current study. Minimum Score: 0. Maximum Score: 24. A higher score means a higher severity of excessive daytime sleepiness.
Epidemiological association of anxiety with CSCR. | At baseline (Month 0), Month 12 and Month 24.
  Generalised Anxiety Disorder (GAD-7) questionnaire: This a validated anxiety scale. Minimum Score: 1. Maximum Score: 21. A higher score means a higher severity of anxiety.
Epidemiological association of depression with CSCR. | At baseline (Month 0), Month 12 and Month 24.
  Patient Health Questionnaire-9 (PHQ-9) questionnaire: This a validated depression scale. Minimum Score: 1. Maximum Score: 27. A higher score means a higher severity of depression.
Epidemiological association of quality of life with CSCR. | At baseline (Month 0), Month 12 and Month 24.
  The National Eye Institute 25-Item Visual Function Questionnaire (NEI-VFQ-25) quality of life questionnaire. Minimum Score: 0. Maximum Score: 100. A higher score means a better vision-targeted health-related quality of life.
Association of single nucleotide polymorphism (SNP) with susceptibility to CSCR | At baseline (Month 0).
  A 10mL blood sample will be drawn from the Participant by venipuncture for DNA sequencing. Odds ratio (OR) (and its 95% confidence interval (CI)) will be calculated to assess the association of the SNP with the susceptibility to CSCR of the Participant.
Number of Participants with serous retinal detachment | At baseline (Month 0), Month 6, Month 12, Month 18 and Month 24.
  Investigators will determine whether serous retinal detachment exists after reviewing the results of functional tests, which include visual acuity and microperimetry, and retinal imaging with non-invasive ultra-widefield colour fundus camera, fundus autofluorescence (FAF) and optical coherence tomography (OCT).

CONTACTS AND LOCATIONS:
Overall Officials: Danny Siu-Chun Ng, FHKAM(Ophth), Principal Investigator — Chinese University of Hong Kong
Locations (3):
- Hong Kong (3):
  - CUHK Eye Centre, Hong Kong
  - Hong Kong Eye Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsai DC, Chen SJ, Huang CC, Chou P, Chung CM, Huang PH, Lin SJ, Chen JW, Chen TJ, Leu HB, Chan WL. Epidemiology of idiopathic central serous chorioretinopathy in Taiwan, 2001-2006: a population-based study. PLoS One. 2013 Jun 24;8(6):e66858. doi: 10.1371/journal.pone.0066858. Print 2013. PMID 23826160
- [Background] Kitzmann AS, Pulido JS, Diehl NN, Hodge DO, Burke JP. The incidence of central serous chorioretinopathy in Olmsted County, Minnesota, 1980-2002. Ophthalmology. 2008 Jan;115(1):169-73. doi: 10.1016/j.ophtha.2007.02.032. PMID 18166410
- [Background] Daruich A, Matet A, Dirani A, Bousquet E, Zhao M, Farman N, Jaisser F, Behar-Cohen F. Central serous chorioretinopathy: Recent findings and new physiopathology hypothesis. Prog Retin Eye Res. 2015 Sep;48:82-118. doi: 10.1016/j.preteyeres.2015.05.003. Epub 2015 May 27. PMID 26026923
- [Background] Chan WM, Lai TY, Lai RY, Liu DT, Lam DS. Half-dose verteporfin photodynamic therapy for acute central serous chorioretinopathy: one-year results of a randomized controlled trial. Ophthalmology. 2008 Oct;115(10):1756-65. doi: 10.1016/j.ophtha.2008.04.014. Epub 2008 Jun 5. PMID 18538401
- [Background] Dansingani KK, Balaratnasingam C, Klufas MA, Sarraf D, Freund KB. Optical Coherence Tomography Angiography of Shallow Irregular Pigment Epithelial Detachments In Pachychoroid Spectrum Disease. Am J Ophthalmol. 2015 Dec;160(6):1243-1254.e2. doi: 10.1016/j.ajo.2015.08.028. Epub 2015 Aug 28. PMID 26319161
- [Background] Ng DS, Bakthavatsalam M, Lai FH, Cheung CY, Cheung GC, Tang FY, Tsang CW, Lai TY, Wong TY, Brelen ME. Classification of Exudative Age-Related Macular Degeneration With Pachyvessels on En Face Swept-Source Optical Coherence Tomography. Invest Ophthalmol Vis Sci. 2017 Feb 1;58(2):1054-1062. doi: 10.1167/iovs.16-20519. PMID 28195603
- [Background] Bakthavatsalam M, Ng DS, Lai FH, Tang FY, Brelen ME, Tsang CW, Lai TY, Cheung CY. Choroidal structures in polypoidal choroidal vasculopathy, neovascular age-related maculopathy, and healthy eyes determined by binarization of swept source optical coherence tomographic images. Graefes Arch Clin Exp Ophthalmol. 2017 May;255(5):935-943. doi: 10.1007/s00417-017-3591-3. Epub 2017 Feb 1. PMID 28150038
- [Background] Lai FH, Ng DS, Bakthavatsalam M, Chan VC, Young AL, Luk FO, Tsang CW, Brelen ME. A Multicenter Study on the Long-term Outcomes of Half-dose Photodynamic Therapy in Chronic Central Serous Chorioretinopathy. Am J Ophthalmol. 2016 Oct;170:91-99. doi: 10.1016/j.ajo.2016.07.026. Epub 2016 Aug 9. PMID 27519561
- [Background] Lai TY, Chan WM, Li H, Lai RY, Liu DT, Lam DS. Safety enhanced photodynamic therapy with half dose verteporfin for chronic central serous chorioretinopathy: a short term pilot study. Br J Ophthalmol. 2006 Jul;90(7):869-74. doi: 10.1136/bjo.2006.090282. Epub 2006 Apr 5. PMID 16597666
- [Background] Chan WM, Lai TY, Lai RY, Tang EW, Liu DT, Lam DS. Safety enhanced photodynamic therapy for chronic central serous chorioretinopathy: one-year results of a prospective study. Retina. 2008 Jan;28(1):85-93. doi: 10.1097/IAE.0b013e318156777f. PMID 18185143
- [Background] van Dijk EHC, Fauser S, Breukink MB, Blanco-Garavito R, Groenewoud JMM, Keunen JEE, Peters PJH, Dijkman G, Souied EH, MacLaren RE, Querques G, Downes SM, Hoyng CB, Boon CJF. Half-Dose Photodynamic Therapy versus High-Density Subthreshold Micropulse Laser Treatment in Patients with Chronic Central Serous Chorioretinopathy: The PLACE Trial. Ophthalmology. 2018 Oct;125(10):1547-1555. doi: 10.1016/j.ophtha.2018.04.021. Epub 2018 Jun 14. PMID 29776672
- [Background] Li WX, Muyese A, Xie ZT, Liu WH, Zhang B. Validity and reliability of the Chinese version of Morningness/Eveningness Questionnaire- 5 items(MEQ-5) in students of technical schools. Chinese Mental Health Journal. 2016; 6: 406-412.